CLINICAL TRIAL: NCT03425825
Title: Treatment Patterns Among Patients With Advanced Small Cell Lung Cancer (SCLC) in Europe
Brief Title: Treatment Patterns in Advanced Small Cell Lung Cancer (SCLC)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-913
Record Dates: First submitted 2017-10-13; First posted 2018-02-08 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer
Keywords: Small Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- LD-SCLC receiving 1st line treatment: patients with LD-SCLC receiving first-line treatment, including potential maintenance treatment
- ED-SCLC receiving 1st line treatment: patients with ED-SCLC receiving first-line treatment, including potential maintenance treatment
- relapsed/refractory receiving 2nd or later-line treatment: relapsed/refractory patients receiving second- or later-line treatment

SUMMARY:
Non-interventional, retrospective study of advanced SCLC patients in 4 European countries (France, Germany, Italy, and United Kingdom [UK]) with the aim to produce evidence across different SCLC treatment lines to characterize the clinical and economic burden of the disease in Europe.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 and 2:

* Patients 18 years of age or older at SCLC diagnosis
* Confirmed diagnosis of SCLC within the patient identification period (between October 2013 and October 2015)
* Initiated on first-line treatment (radiotherapy and/or chemotherapy) for their SCLC
* Full oncology medical history for the mandatory variables of the study available in the participating center from day of diagnosis until the end of follow-up or death (whichever occurs first)
* Signed informed consent (where required as per local requirements)

Cohort 3:

* Patients 18 years of age or older at SCLC diagnosis
* Confirmed diagnosis of SCLC not earlier than October 2013
* Initiated on second-line treatment due to relapse after first-line therapy not later than August 2016
* Full oncology medical history for the mandatory variables of the study available in the participating center from day of diagnosis until the end of follow-up or death (whichever occurs first)
* Signed informed consent (where required as per local requirements)

Exclusion Criteria:

* Participants with previous malignancies (except non-melanoma skin cancers, and in situ cancers such as the following: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to first treatment and no additional therapy is required or anticipated to be required during the study period.

Other Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced SCLC patients in 4 European countries (France, Germany, Italy, and United Kingdom [UK]).
Sampling Method: Non-Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Distribution of Patient Demographic Characteristics | At baseline
  Characteristics include:
  Age/month and year of birth Gender Ethnicity Weight Height Smoking status Alcohol consumption Other relevant risk factors
Distribution of Patient Clinical Characteristics in Relapsed/refractory patients receiving second- or later-line treatment | At baseline
  Characteristics include:
  Relevant comorbidities Laboratory parameters Date of initial diagnosis Staging using the VALG system Histology ECOG Performance status Tumor status Symptoms
Distribution of Patient Clinical Characteristics in patients with LD-SCLC | At baseline
  Characteristics include:
  Relevant comorbidities Laboratory parameters Date of initial diagnosis Staging using the VALG system Histology ECOG Performance status Tumor status Symptoms
Distribution of Patient Clinical Characteristics in patients with ED-SCLC | At baseline
  Characteristics include:
  Relevant comorbidities Laboratory parameters Date of initial diagnosis Staging using the VALG system Histology ECOG Performance status Tumor status Symptoms
Distribution of treatment patterns in patients with ED-SCLC | Approximately 44 months
  Details on patients prior treatment Patterns will be summarized using descriptive statistics
Distribution of treatment patterns in patients with LD-SCLC | Approximately 44 months
  Details on patients prior treatment Patterns will be summarized using descriptive statistics
Distribution of treatment patterns in Relapsed/refractory patients receiving second- or later-line treatment | Approximately 44 months
  Details on patients prior treatment Patterns will be summarized using descriptive statistics

SECONDARY OUTCOMES:
Composite of SCLC-related healthcare resource utilization (HCRU) | Approximately 44 months
  HCRU will include hospitalizations, emergency visits, outpatient visits, treatments received (including treatments prescribed to manage AEs), diagnostic tests and procedures, surgery, and ancillary services.
Overall survival (OS) | Approximately 44 months
Progression-free survival (PFS) | Approximately 44 months
Objective response rate (ORR) | Approximately 44 months
Mortality rate | Approximately 44 months
Treatment-related adverse events (AEs) leading to discontinuation | Approximately 44 months
Incidence of surgery as cancer-directed therapy | Approximately 44 months
  To describe the use of surgery in the management of LD-SCLC and ED-SCLC patients having relapsed
Incidence of radiation therapy as cancer-directed therapy | Approximately 44 months
  To describe the use of radiation therapy in the management of LD-SCLC and ED-SCLC patients having relapsed
Incidence of best supportive care (BSC) | Approximately 44 months
  To describe the use of best supportive care (BSC) in the management of LD-SCLC and ED-SCLC patients having relapsed
Incidence of palliative care | Approximately 44 months
  To describe the use of palliative care in the management of LD-SCLC and ED-SCLC patients having relapsed

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution, Barcelona, Spain
- Local Institution, London, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm